CLINICAL TRIAL: NCT03324360
Title: The Feasibility and Role of Hyperpolarized 13C-Pyruvate MR Spectroscopy in Monitoring Patients With Intracranial Metastasis Treated With Stereotactic Radiosurgery (SRS)
Brief Title: Role of Hyperpolarized 13C-Pyruvate MR Spectroscopy in Patients With Intracranial Metastasis Treated With (SRS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 333-2014
Record Dates: First submitted 2017-10-04; First posted 2017-10-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Participants Part I (Experimental): A MRI with injection of hyperpolarized 13C pyruvate.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate
- Intracranial Metastasis Part II (Experimental): MRI with injection of hyperpolarized 13C pyruvate prior to radiation treatment.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate
- Intracranial Metastasis Part III (Experimental): MRI with injection of hyperpolarized 13C pyruvate prior to radiation treatment. MRI with injection of hyperpolarized 13C pyruvate following radiation treatment.
  MRI with injection of hyperpolarized 13C pyruvate following radiation treatment if adverse radiation effect is identified on post-SRS follow-up images.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — MRI with Hyperpolarized 13C-Pyruvate Injection

SUMMARY:
Upwards of 40% of cancer patients will develop brain metastases during their illness, most of which become symptomatic. The burden of brain metastases impacts the quality and length of survival. Thus the management of brain metastases is a significant health care problem. Standard treatment options include stereotactic radiosurgery and/or whole brain radiation. There is a great interest in studying the association between the functional characteristics of tumors - such as tumour hypoxia and lactate accumulation - and clinical outcomes in order to guide management. These characteristics may predict future tumor behavior and stratify risk of therapy failure. Hyperpolarized 13C MR imaging is a novel functional imaging technique that uses 13C-labeled molecules, such as pyruvate, and MRS to image in vivo tissue metabolism.

There is significant clinical heterogeneity in patients with brain metastasis due to differences in underlying tumour biology. Biochemical differences in tumour metabolism have been shown to correlate with response to therapy. While the significance of tissue hypoxia for radiosensitivity has been established for years, the impact of lactate accumulation on radiosensitivity has only recently been recognized. Studies have shown that tissue lactate levels correlate with radioresistance in several human tumours. Hyperpolarized 13C pyruvate MRS has been shown in numerous pre-clinical studies and a recent clinical study to have great potential as a metabolic imaging tool. Our study seeks to establish the role of hyperpolarized 13C MRS in characterizing the metabolic features of intracranial metastasis. The results of this study will provide insight into intracranial metastatic disease signatures with MR spectroscopy and determine if there is added benefit for incorporation of this new technique into future clinical MRI protocols. If the technique can accurately differentiate between aggressive and indolent tumours based on MR spectroscopic patterns, hyperpolarized 13C MRS may have wide-ranging utility in the future. In the era of personalized medicine, the ability of imaging tests to predict response to therapy would open the door for individualized treatment options specific to each patient's disease biology.

DETAILED DESCRIPTION:
This is a pilot prospective, single-institution study in both control participants, control participants with mild cognitive impairment and Alzheimer's disease and participants with evidence of intracranial metastases who will be planned for brain radiation therapy. Control participant accrual will be done through advertisements. For control participants with mild cognitive impairment, Alzheimer's disease and intracranial metastatic disease screening and accrual will be completed by a member of the participant's Circle of Care. Clinical procedures will be completed at Sunnybrook Health Sciences Centre (SHSC) by the study's Qualified Investigator or medical designate. Eligible control participants must meet the study's inclusion and exclusion criteria and MRI eligibility. Intracranial metastatic participants must meet the study's inclusion and exclusion criteria, MRI eligibility will be undergoing radiation therapy (stereotactic radiotherapy).

The study will be divided into three parts:

Part I (Controls)

* Population: up to 146 study participants, ≥18 years of age
* Each participant in Groups A to G and J and K will undergo a single MRI sequence with a single hyperpolarized 13C pyruvate injection. Participants in group H, I, and M will undergo MRI sequences with two consecutive injections of hyperpolarized 13C pyruvate. The scans are expected to be of approximately 60 to 75 minutes in length.

Group A: up to 6 participants ≥ 18 years of age. Group B: up to 10 male participants between the age of 18-39 Group C: up to 10 female participants between the age of 18-39 Group D: up to 10 male participants between the age of 40-59 Group E: up to 10 female participants between the age of 40-59 Group F: up to 10 male participants ≥ 60 years of age Group G: up to 10 female participants ≥ 60 years of age Group H: up to 10 male or female participants ≥ 18 years of age Group I: up to 10 male or female participants ≥ 18 years of age Group J: up to 10 male or female participants ≥ 60 years of age with Mild Cognitive Impairment Group K: up to 10 male or female participants ≥ 60 years of age with Alzheimer's disease Group L: up to 10 male or female participants ≥18 years of age Group M: up to 30 male or female participants ≥18 years of age

Part II

* Population: up to 100 study participants from the Odette Cancer Centre, ≥18 years of age with demonstrated intracranial metastasis on imaging (CT or MRI), who have been referred to clinic for radiotherapy consideration.
* Procedure: Each participant will undergo additional MRI sequences (hyperpolarized 13C pyruvate MRS) with an additional length of approximately 30-60 minutes that will be performed on the day of or in advance of the participant's routine radiation planning scan prior to radiation treatment. No extra visits to the hospital, beyond routine clinical care, are anticipated.

Part III

* Population: up to 30 study participants from the Odette Cancer Centre, ≥18 years of age with demonstrated intracranial metastasis on imaging (CT or MRI), who have been referred to clinic for radiotherapy consideration.
* Procedure: Each participant will undergo additional MRI sequences (hyperpolarized 13C pyruvate MRS) with an additional length of approximately 30-60 minutes that will be performed on the day of or in advance of the participant's routine radiation planning scan prior to radiation treatment, or following treatment. In addition, if an adverse radiation effect is identified on post-SRS follow-up images by the qualified investigator, each participant will undergo non-routine MRI scans with a length of approximately 60-90 minutes. Participants who do not receive a pre-SRS hyperpolarized 13C pyruvate MRS scan, but that present with an ARE post-SRS, are also included in this population. The quantity of follow-up scans will be as deemed necessary by the qualified investigator.

ELIGIBILITY:
Inclusion Criteria:

Part I (Controls) Group A

* Participants of all ethnic groups/race categories (≥18yrs old)
* Informed consent Group B
* Male participants of all ethnic groups/race categories (between the age of 18-39)
* Informed consent Group C
* Female participants of all ethnic groups/race categories (between the age of 18-39)
* Informed consent Group D
* Male participants of all ethnic groups/race categories (between the age of 40-59)
* Informed consent Group E
* Female participants of all ethnic groups/race categories (between the age of 40-59)
* Informed consent Group F
* Male participants of all ethnic groups/race categories (≥60 yrs old)
* Informed consent Group G
* Female participants of all ethnic groups/race categories (≥60 yrs old)
* Informed consent Group H and I
* Male or female participants of all ethnic groups/race categories (≥18 yrs old)
* Informed consent Group J
* Male or female participants of all ethnic groups/race categories (≥60 yrs old)
* Informed consent
* Diagnosed with mild cognitive impairment Group K
* Male or female participants of all ethnic groups/race categories (≥60 yrs old)
* Informed consent
* Diagnosed with mild Alzheimer's disease Group L
* Male or female participants of all ethnic groups/race categories (≥18 years of age)
* Informed consent Group M
* Male or female participants of all ethnic groups/race categories (≥18 years of age)
* Informed consent

Part II & III

* Adult participants of all ethnic groups/race categories (age ≥18 yrs old)
* Radiographic diagnosis of brain metastases and pathological confirmation of a solid cancer primary
* Metastatic brain tumor amenable to Stereotactic radiosurgery or radiotherapy
* Participants on dexamethasone must be on a stable dose at the time of baseline MRI and 1-5 days post-SRS MRI
* Estimated survival more than 6 months
* Informed consent

Exclusion Criteria:

* Prior brain radiotherapy for the specific index or lesion to be imaged in the study
* For groups B to I, L, and M only: Montreal Cognitive Assessment (MoCA) score <26
* The participant will also be asked to complete the standard MRI safety screening questionnaire, prior to their research scan and participation in the study.
* Contraindications to MRI including:
* Participants weighing >136 kg (weight limit for the scanner tables)
* Participants with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI.
* Pregnant
* Claustrophobia to the extent that the participant cannot stay in the MRI for 45-60 minutes
* Known adverse reactions to the contrast agent Gd-DTPA
* Inability to lie still for 45-60 minutes
* Participants with a high risk factor for nephrogenic systemic fibrosis (NFS).
* Participant declines the procedure or further procedures;
* Participant is not well enough to undergo MRI scanning;
* Participant is unable to complete the MRI procedure for any reason or is non-compliant with MRI requirements.
* For groups J and K, a <1 lacunar infarct or any cortical subcortical infarct or moderate to severe white matter disease
* For groups J and K, any other structural brain lesion that could affect cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Is an MRI image produced? Y/N? | ~30-60 minutes of MRI time.
  To demonstrate the first 13C-metabolic images of the human brain, alone with the required hardware and data acquisition methods.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No